CLINICAL TRIAL: NCT04438824
Title: A Phase II Study of CDK4/6 Inhibition (Palbociclib) Combined With PD-1 Blockade (INCMGA00012) in Patients With Advanced Well-differentiated Dedifferentiated Liposarcoma
Brief Title: Palbociclib and INCMGA00012 in People With Advanced Liposarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-062; R01FD007528-01 (FDA)
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Well-differentiated/Dedifferentiated Liposarcoma
Keywords: Palbociclib; INCMGA00012; 20-062
MeSH Terms: conditions — Liposarcoma | interventions — palbociclib

STUDY DESIGN:
Intervention Model Description: This is a phase II study of palbociclib plus INCMGA00012 in patients with advanced WD/DD liposarcoma.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Palbociclib and INCMGA00012 (Experimental): Initial design (safety lead-in and expansion): One treatment cycle will consist of 28 days. Patients in both study phases will start palbociclib on Day 1 and INCMGA00012 on day 15 (+/- 7 days) of each cycle at the following dose schedule: INCMGA00012: 500 mg IV (flat dose) q28 days Palbociclib: 125 mg PO daily for 21 days, followed by 7 days off, q28 days Palbociclib will be taken on Day 1 of each cycle for 21 consecutive days followed by 7 days off (days 22-28 of each Cycle). INCMGA00012 will be administered on Day 15 of (+/- 7 days) each cycle and repeat every 28 days.(No longer using this)
  Amended design (Expansion only): One treatment cycle will consist of 28 days. Patients in both study phases will start palbociclib and INCMGA00012 on day 1 of each cycle: 500 mg IV (flat dose) of INCMGA00012 will be administered q28 days concurrently with palbociclib 125 mg PO daily for 21 days, followed by 7 days off, q28 days.
  Interventions: Drug: INCMGA00012; Drug: Palbociclib

INTERVENTIONS:
Drug: INCMGA00012 — INCMGA00012: 500 mg IV (flat dose) q28 days (+/- 7 days in each cycle)
Drug: Palbociclib — Palbociclib:125 mg PO daily for 21 days, followed by 7 days off, q28 days

SUMMARY:
The researchers are doing this study to find out whether combining the study drugs palbociclib and INCMGA00012 is an effective and safe treatment for advanced liposarcoma.

"Funding Source - FDA OOPD"

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of metastatic or unresectable WD/DD liposarcoma. DD liposarcoma must be present. Unresectable is defined as if the primary tumor a) cannot be safely removed surgically or b) would benefit from systemic therapy prior to a surgical approach
* Measurable disease by RECIST 1.1

  a. Target lesions must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to enrollment
* Age ≥ 18 years
* ECOG performance status 0 or 1
* Adequate organ and marrow function as defined below (ULN indicates institutional upper limit of normal):

  1. Absolute neutrophil count ≥ 1.5 x 109/L
  2. Hemoglobin ≥ 8.0 g/dL
  3. WBC ≥ 3.0 x 109/L
  4. Platelets ≥ 100 x 109/L
  5. ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN. Except patients with Gilbert's disease (≤3x ULN)
  6. AST (SGOT) /ALT (SGPT) ≤ 3 x institutional ULN
  7. Creatinine Clearance > 30 mL/min (calculated by Cockcroft-Gault method)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) during the trial period through at least 120 days after the last dose of study treatment.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow tablets or capsules
* Patients with brain metastasis that have been treated with definitive surgery or radiation, and have been clinically stable for 3 months are eligible

Exclusion Criteria:

* Patients who have not recovered from clinically significant adverse events of prior therapy to ≤ NCI CTCAE v5 Grade 1, except alopecia and stable neuropathy, which must have resolved to Grade ≤ 2 or baseline.
* Patients receiving any other investigational agents.
* Patients who have received prior treatment with a selective CDK4 inhibitor or an anti-PD-1/PD-L1 agent
* Uncontrolled intercurrent illness including, but not limited to, known ongoing or active infection, including uncontrolled HIV, active hepatitis B or C, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmias, psychiatric illness/social situations that would limit compliance with study requirements, clinically significant interstitial lung disease or active noninfectious pneumonitis, or active infection requiring systemic therapy

  1. Patients with a CD4+ count of > 300 and an undetectable viral load who are currently on HAART are eligible for inclusion
  2. Patients with NYHA class III or IV congestive heart failure within 6 months of study treatment will be excluded
* Pregnant women and women who are breast-feeding.
* History or evidence of symptomatic autoimmune disease in past 2 years prior to enrollment.

  a. Replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease
* Prolonged QTcF > 450 ms for men and > 470 ms for women at Screening.
* Patients who have received a live vaccine within 30 days of the start date of the planned study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines are live attenuated vaccines, and are not allowed
* Radiation therapy within 2 weeks prior to study Day 1
* Prior organ transplantation including allogenic stem-cell transplantation
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v 5 Grade ≥ 3)
* Patients who require concomitant use of medications that strongly induce or inhibit CYP3A (per section 15.0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
confirm the recommended phase two dose (RP2D | within 6 weeks of treatment
  DLTs will be assess within the first 6 weeks of the treatment combination . DLT definitions are described in section 15.4, and will be defined using NCI CTCAE v 5.0. If ≤ 1 patient out of 6 has a dose-limiting toxicity, the dosing used in the safety lead-in phase will be declared the recommended phase 2 dose. If ≥ 2 of 6 patients in the safety lead-in experience a DLT, study treatment will be halted and no further patients will be enrolled. If the study is resumed with an alternative dosing schema, a new safety lead-in phase will be completed with the new dosing regimen
best overall response rate (Phase II) | by 48 weeks
  defined by RECIST 1.1

SECONDARY OUTCOMES:
Safety | 2 years
  Safety will be assessed using CTCAE v 5.0 to define that adverse event profile of the treatment combination and safety events will be tabulated.
overall response rate | 48 weeks
  as defined by irRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D'Angelo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT04438824/ICF_000.pdf